CLINICAL TRIAL: NCT02392936
Title: Evaluation of Peri-operative Risk Factors for Surgery Site Infection in Cardiac Surgery
Acronym: PRISCCA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Paul-Henri WICKY, Anesthésiste-Réanimateur, Centre Hospitalier Universitaire de Besancon
Other Study IDs: CHU Besancon
Record Dates: First submitted 2015-03-04; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Surgical Site Infection
Keywords: according to the definition of the Comité Technique des Infections Nosocomiales et Liées aux Soins (2007)
MeSH Terms: conditions — Surgical Wound Infection | interventions — Sternotomy; Coronary Artery Bypass; Nuclear Receptor Subfamily 4, Group A, Member 2; Appointments and Schedules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood samples during and after intervention, for routine tests, and eventually dosing plasmatic concentration of the antibiotic administered for prophylaxis. Microbiological analyses concerning wound and blood samples.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sternotomy for coronary artery bypass graft, valvuloplasty, aortic surgery or combined procedures, under extracorporeal circulation or not, in emergency or scheduled.

SUMMARY:
There is a recent increase in incidence of surgical site infection after cardiac surgery in our hospital, in spite of specific measures taken concerning some aspects of the surgical procedures, targeting a better control of the classically known major risk factors of infections, in routine procedures involving a sternotomy such as coronary artery bypass graft, valvuloplasty, aortic surgery, or combined procedures.

The first objective of this monocentric prospective cohort study, is to evaluate underestimated specific risk factors of surgical site infection, during the perioperative period, for patients undergoing cardiac surgery with sternotomy.

Secondly, to estimate the specific risk associated with each class or micro-organisms responsible, and their profile of resistance.

The outcomes concern the occurrence of a surgical site infection diagnosed by the surgeon in charge of the patient, one month and three months after surgery; it may concern the pre operative period, the procedure itself, or the early post operative period, characterized by a high density of cares, or even the late rehabilitation, after discharge of the surgical unit.

Secondary outcome evaluate the profile of agents identified regarding the susceptibility of the prophylaxis recommended to prevent wound infection; it may suggest that an adequate antibiotic prophylaxis is often insufficient to take into account the responsible agents, and that decolonisation is not always that helpful, in view of emerging cases of failure due to developing resistance.

Considering the low incidence of that type of complication, the investigators estimated that a period of two years might be necessary to include a sufficient number of patient, at least one thousand, in order to find a dozen of factors that might be significantly associated with an increased risk of surgical site infection.

The evaluation is permitted by the collaboration between the anesthesiologists, surgeons, intensivists, hygienists, all along the presence of the patient in the department, until discharge out of the hospital and after readmission eventually for infectious complication.

DETAILED DESCRIPTION:
Surgical site infection following cardiac surgery is source of a significant morbidity and mortality. It may occur in patients who present preexisting fragilizing underlying conditions, and who suffer a major surgical traumatism, considering the sternotomy, the presence of an eventual extracorporeal circulation, the bleeding risk associated to the procedure, hypothermia, etc.

Many risk factors have already been studied, and might be targeted by prevented measures.

Some of them concern the pre-operative period, related to the patient's underlying conditions, the disinfection and eventual decolonisation of the patients; some concern the procedure intrinsically, according to the surgical technique preferred; an important role may be accorded to the post-operative period, during which a high density of care might be responsible of an eventual contamination, recolonisation, or fragilisation of the patients, thus making them more susceptible to infection.

Despite the control of the modifiable risk factors and the application of preventive measures, we are facing a progressive increasing in surgical site infection since a few months.

We aim to prospectively and exhaustively evaluate all the risk factors that can play a role before, during or after the surgical period, in the routine procedures involving a sternotomy, including coronary artery bypass graft, valvuloplasty (except for endocarditis), thoracic aortic surgery, and combined procedures, without considering the degree of emergency, the presence of an extracorporeal membrane, in every major adult admitted in the department of cardiothoracic surgery.

Those events can be related to the contemporary increased activity in the department of cardiothoracic surgery. This hypothesis was advanced as an explanation, but the growing number of patients operated during the last months couldn't be the only factor responsible of the post-operative infectious complications. Moreover, microbiological epidemiology does not simply allow a single targeted preventive strategy because there is no particular agent responsible of these infections, and the bacterial populations are globally comparable to the classical ones identified in this type of surgery. It is including of large majority of gram positive cocci, essentially Staphylococcus aureus (in which we find a quasi absence of methicillin-resistance) and epidermis, and a significant prevalence of gram negative bacilli. So there is no evidence of an epidemic recrudescence linked to a specific microbiological element that could be easily identified.

Nevertheless, the recommended prophylaxis deserve to be reconsidered, regarding the overall emergence in every class of microbial agents, which constitute a real problem that have to face each intensive care unit; thus, it seems logical to consider that the same protocol applied during several years may lose in efficacy while the epidemiology of resistance is in constant and accelerating evolution. So the microbial agents could be identical as those classically identified, so may not their susceptibility. At least, we might consider an eventual modification of our choices in which prophylaxis should be administered.

The evaluation starts preoperatively after information of the eligible patients, at the admission in the cardiothoracic department, while it can also be initiated during the preoperative anesthaesic evaluation. In all case, a moment before admission in operating room should be dedicated by a resident in surgery or anesthesiolgy to recense the pre existing conditions.

Then the time of the procedure may involve different actors (perfusionist, all member of the anesthesiologic team, surgeons) to examine each step of the procedure, pre-established on a checklist to which every one has access (informed file for each patient who enter the operating room).

After surgery, the cares occur in a dedicated unit as long as the patient's status justify intensive monitoring, often invasive, and eventual appropriate suppliance mediated by drugs or devices according to intensivist praticians in charge, surgeon or anesthesiologist, the procedure and the patient's tolerance.

As early as possible, the discharge of this unit is decided to pursuit in a conventional sector, where the patient is in charge of the surgical staff only, with a more moderate surveillance but to permit an early rehabilitation, before discharge of the hospital, towards a rehabilitation facility, and then return at home.

The follow-up is commonly accomplished by all the actors taking part in the operating room, and after in the intensive care unit. But during hospitalisation or after discharge, it is the surgeons' role to diagnose and declare to hygienists all the infectious complications that might be considered as surgical site infection. In case of re-admission for complications, the hygienist staff should also receive such a declaration.

In order to collect exhaustively all the interesting variables before, during and after surgery, for a period potentially prolonged until 3months, one member of the anesthesiologist staff is in charge to audit the follow-up in every care unit inside hospital from admission until discharge, and also after check if an eventual event occurred, with the hygienists informed of that event.

An ancillary study might next be conducted, in order to evaluate the pharmacokinetic of antibiotic prophylaxis for patient under extracorporeal circulation. It might eventually study the modality of continuous administration over a prolonged time during surgery; it might include blood samples during procedure and immediately after for repeated antibiotic dosages.

Sites were blood sample is taken can be extracorporeal circulation or catheter used for routine monitoring, such as radial artery catheter, for invasive blood pressure monitoring, which is a constant mean of surveillance peroperatively and after surgery in intensive care unit.

So this procedure does not implicate further invasive manipulations that are not already in part of the routine standard cares.

ELIGIBILITY:
Inclusion Criteria:

* patient aged more than 18 yards old,
* sternotomy for one of the following procedures : coronary artery bypass, valvuloplasty, aortic surgery, combination of the mentioned interventions.
* without considering the degree on emergency and the presence of extra corporeal circulation.

Exclusion Criteria:

* patient under age or 18years old.
* patient not informed.
* surgical revision in case of suspicion of infection, haemorragic complication, suspicion of myocardial infarction.
* endocarditis indicating a valvuloplasty procedure.
* patient who underwent orthopedic surgery with prothetic material, within the 12 months preceeding cardiac procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient undergoing a cardiac procedure with sternotomy, including coronary artery bypass, " , aortic surgery, or combined procedures, scheduled or on emergency, under extracorporeal circulation or not.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Surgical Site infection | 30 days after surgery
  Diagnostic made by the surgeon in charge of the patient, according to the criterias suggested by the CTINLS, on clinical or paraclinical elements.
  The occurrence during the first month may point out a potential interest of an intervention on a short term period (during and after surgery), concerning the cares administered inside the department of cardiothoracic surgery.
Surgical Site Infection | 90 days after surgery
  Diagnostic made by the surgeon in charge of the patient, according to the criterias suggested by the CTINLS, on clinical or paraclinical elements.
  The occurence of a delayed diagnosis may suggest a late infection, involving an intervention during and after the rehabiliation, outside the departement of cardiothoracic surgery.
  Some elements may concern the surgical period, but my be revealed several weeks after the discharge of the patient.

SECONDARY OUTCOMES:
Bacterial Phenotype regarding the molecule administered as prophylaxis or decontamination preoperatively or during the procedure. | 30 days after surgery
  The bacterial agent, causing the surgical site infection, susceptibility or resistance towards the antibiotic prophylaxis and the decontamination agents.
  Accurately, the susceptibility to mupirocin, cefuroxime, and vancomycin can vary and explain an early and agressive developement in the wound site.
Bacterial Phenotype regarding the molecule administered as prophylaxis or decontamination preoperatively or during the procedure. | 90 days after surgery
  The bacterial agent, causing the surgical site infection, susceptibility or resistance towards the antibiotic prophylaxis and the decontamination agents.
  Accurately, the susceptibility to mupirocin, cefuroxime, and vancomycin can vary and allow a low and delayed developement in the wound region.